CLINICAL TRIAL: NCT01826630
Title: A Double-Blind Pilot Study To Assess The Feasibility of a Larger Study to Assess The Efficacy of A Novel Gel Wash Cleanser Formulated With Sodium Hypochlorite To Reduce Skin Fauna In Patients With Chronic Hand Dermatitis/Atopic Dermatitis.
Brief Title: A Study to Assess CLn® BodyWash for Reducing Skin Fauna in Patients With Hand Eczema
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: Shari L Hand (Industry)
Collaborators: TopMD Skin Care, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Shari L Hand, Clinical Research Director, TopMD Skin Care, Inc.
Organization: TopMD Skin Care, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CLN 2012H0327
Record Dates: First submitted 2013-02-20; First posted 2013-04-08 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2014-11

CONDITIONS: Eczema; Hand Eczema; Atopic Dermatitis
Keywords: CLn Body Wash; CLn BodyWash
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CLn BodyWash (Active Comparator): CLn BodyWash will be used to wash hands of patients with Hand Atopic Dermatitis
  Interventions: Other: CLn BodyWash
- Cetaphil Daily Facial Cleanser (Active Comparator): Cetaphil Daily Facial Cleanser will be used to wash hands of patients with Hand Atopic Dermatitis
  Interventions: Other: Cetaphil Daily Facial Cleanser

INTERVENTIONS:
Other: CLn BodyWash — Comparing two washes to determine change in bacterial load.
  Arms: CLn BodyWash
Other: Cetaphil Daily Facial Cleanser — Comparing two washes to determine change in bacterial load.
  Other Names: Cetaphil Daily Facial
  Arms: Cetaphil Daily Facial Cleanser

SUMMARY:
The primary objective of this protocol is to acquire pilot data for a larger study to test the following hypothesis: Treatment of the hands of patients with chronic hand dermatitis/atopic dermatitis with CLn BodyWash, a novel gel wash cleanser currently marketed as a cosmetic product containing a dilute concentration of less than 0.01% sodium hypochlorite and less than 0.005% concentration as it is lathered, will result in a statistically significant reduction in the number of skin fauna present on the hands of these patients compared to treatment of such patients with traditional wash used clinically such as Cetaphil Daily Facial Cleanser.

DETAILED DESCRIPTION:
Patients with Hand Eczema will be asked to wash with either a CLn BodyWash or Cetaphil Daily Facial Cleanser. Patients and study staff will be blinded. Hand swabs will be done prior to the wash and after 20 minutes. The average time spent in the study for each patient should be less than 2 hours unless an Adverse Event occurs.

ELIGIBILITY:
Inclusion Criteria:

* Seen by an OSU Dermatology provider at OSU Dermatology East after the date of approval of this protocol
* Ability to provide informed consent, or parent or legal guardian capable of providing consent for child or mentally handicapped individuals
* Willingness to participate in a research study.
* Diagnosis of chronic hand dermatitis

Exclusion Criteria:

* Inability to provide informed consent
* Allergy to any of the treatments used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Amount of Skin Fauna | one wash
  Mean Decrease in Fauna after Washing with either CLn BodyWash or Cetaphil Daily Facial Cleanser.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Gahanna, Ohio, United States